CLINICAL TRIAL: NCT05167682
Title: Patient Empowerment for Major Surgery Preparation @ Home
Acronym: PAPRIKA
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: Department of General, Visceral, Tumor and Transplant Surgery, University Hospital Of Cologne (Unknown); Centre for Prevention and Rehabilitation, University Hospital Cologne (Unknown); Department of Endocrinology, Diabetology and Preventive Medicine (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Paul Brinkkoetter, Prof. MD, Consultant in Nephrology, University Hospital of Cologne
Other Study IDs: V02-20012021
Record Dates: First submitted 2021-07-22; First posted 2021-12-22 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Transthoracic Esophagectomy
Keywords: Transthoracic esophagectomy; Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prehabilitation: 25 patients scheduled for tumor-esophagectomy (Ivor-Lewis) who are capable and have given consent to participate in a smartphone-based prehabilitation program.
  Interventions: Other: Prehabilitation program
- Historical Cohort: Patients ≥ 65 years of age who have undergone tumor-related esophagectomy at the University Hospital of Cologne between 05/2016 and 04/2020, who have not participated in any form of prehabilitation procedures

INTERVENTIONS:
Other: Prehabilitation program — Patient will be asked to follow to catalog of procedures till surgery. Procedures catalog contains behavioral changes, physical training, nutritional counseling, conditioning of pulmonary function and optimization of drug of underlying diseases.
  Groups: Prehabilitation

SUMMARY:
The PAPRIKA project is a feasibility study with duration of 10 months. The aim of the study is to recruit 25 patients over the age of 65 who will undergo tumor-related esophagectomy and will follow a prehabilitation program to prevent postoperative complications and improve patient-centric complications and patient-centered outcomes.

After determination of the oncologic treatment plan in the tumor board and functional assessment, patient will undergo an interdisciplinary assessment , which will be performed by the PAPRIKA team consisting of physiotherapists, internists/geriatricians, speech and occupational therapists, nutritionists and surgeons.

On the basis of this interdisciplinary assessment an individualized catalog of procedures will be created. Patient have to follow to this catalog of procedures until surgery. Procedures catalog contains behavioral changes, physical training, nutritional counseling, conditioning of pulmonary function and optimization of drug treatment of underlying diseases.

The individual treatments will be weekly reevaluated and if necessary the procedures will be adjusted by treatment teams.

The prehabilitation procedures will be communicated with the patient via a smartphone app, which is specially developed for the prehabilitation program. The implementation will be documented.

The primary aim of this study is to evaluate the compliance of the patients regarding to the prescribed procedures and the use of the smartphone app (feasibility).

As secondary aim postoperative outcome will be compared with the results of a historical cohort for quality control.

ELIGIBILITY:
Inclusion Criteria

* Patients ,undergoing transthoracic esophagectomy (Ivor Lewis), in ≥ 4 weeks
* Age >65 years
* American Society of Anaesthesiologists - Score: 2-3
* Ability to give informed consent
* Written informed consent

Exclusion Criteria:

* Planned operation in less than 4 weeks after enrollment
* Urgent surgery indication
* Patients with good to excellent general and nutritional condition (0 points in the pre-screening of the modified NRS OR 1 point in the pre-screening and <2 points in the main screening).
* Patients deemed by the PAPRIKA team to be physically or mentally incapable of completing the exercise program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Male and female subjects with planned transthoracic esophagectomy in more than 4 weeks
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Compliance of patients as feasibility of prehabilitation program | 90 days after surgery
  Percentage of patients will be assessed, who have successfully completed all study visits and have installed and used the smart phone app at least once

SECONDARY OUTCOMES:
Postoperative outcome | 90 days after surgery
  Postoperative outcome will be measured with occurrence of postoperative and patient-centric complications.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Schröder, Prof., Study Chair — Department of General, Visceral and Transplantational Surgery, University Hospital of Cologne; Paul Brinkkötter, Prof., Principal Investigator — Department of Internal Medicine II, University Hospital of Cologne; Linus Völker, MD, Principal Investigator — Department of Internal Medicine II, University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No